CLINICAL TRIAL: NCT07379333
Title: A Multicenter, Randomized, Double-blind, Phase 3 Study to Evaluate Efficacy and Safety of HM11260C in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin and Dapagliflozin
Brief Title: A Study to Evaluate Efficacy and Safety of HM11260C in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin and Dapagliflozin
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-GLOW-301
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HM11260C (Experimental): Weekly administration by subcutaneous injection
  Interventions: Drug: HM11260C
- Placebo (Placebo Comparator): Weekly administration by subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HM11260C — Test drug
  Arms: HM11260C
Drug: Placebo — Placebo drug
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, phase 3 study to evaluate efficacy and safety of HM11260C in patients with type 2 diabetes mellitus inadequately controlled with metformin and dapagliflozin

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults aged 19 years or older
* 2. Diagnosed with type 2 diabetes
* 3. HbA1c level 7.0% ≤ HbA1c ≤ 10.0%
* 4. Stable administration of metformin (≥1,000 mg/day) and dapagliflozin (10 mg/day) without any change in dosage or formulation for at least 8 weeks prior to Visit 1
* 5. 20 kg/m2 ≤ BMI ≤ 45 kg/m2
* 6. Agree to the recommended exercise and diet regimen during this clinical trial

Exclusion Criteria:

* 1. Patients with a history of allergy or resistance to the investigational drug or background therapy
* 2. Patients diagnosed with a type of diabetes other than type 2 diabetes
* 3. Patients with uncontrolled severe diabetic complications
* 4. Patients with a history of acute or chronic metabolic acidosis, including lactic acidosis or diabetic ketoacidosis.
* 5. Patients with a history of diabetic coma or precoma
* 6. Those with a history of severe hypoglycemia
* 7. Those whose weight change > 5 kg
* 8. History of gastrointestinal disease or surgery
* 9. History of bariatric surgery
* 10. History of gallbladder disease
* 11. History of a disease that could affect the interpretation of HbA1c
* 12. History of acute or chronic pancreatitis or pancreatectomy
* 13. History (including family history) of medullary thyroid cancer (MTC) or multiple endocrine neoplasia (MEN2).
* 14. Uncontrolled hypertension
* 15. Severe infections or severe trauma
* 16. Malnutrition, starvation, or debility, as determined by the investigator.
* 17. Pituitary or adrenal insufficiency.
* 18. Tissue hypoxia, such as respiratory failure or shock.
* 19. History of alcoholism or drug abuse
* 20. History of malignant tumors
* 21. Heart failure, Ischemic heart disease, Severe cerebrovascular disease, TIA
* 22. Patients with one of the following clinical laboratory test results : Amylase or Lipase > 3 X ULN / FPG > 270 mg/dL
* 23. Patients with severe hepatic impairment or one of the following laboratory test results : AST or ALT > 3 X ULN / Total bilirubin > 1.5 X ULN
* 24. Patients with moderate or severe renal impairment
* 25. History of Diabetic medications or weight-loss medications
* 26. Those who have participated in another clinical trial and received investigational drugs within 30 days
* 27. Pregnant or lactating women, or women of childbearing potential
* 28. Women of childbearing potential and men who do not consent to the use of the following contraceptive methods
* 29. Considered by investigator as not appropriate to participate in the clinical study with other reason.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c at 36 weeks compared to baseline | baseline, 36 weeks

SECONDARY OUTCOMES:
Change from baseline in HbA1c at Week 24 | baseline, 24 weeks
Proportion of subjects achieving HbA1c <7.0% at Weeks 24 and 36 | 24, 36 weeks
Proportion of subjects achieving HbA1c <6.5% at Weeks 24 and 36 | 24, 36 weeks
Change from baseline in FPG at Weeks 24 and 36 | baseline, 24, 36 weeks
Proportion of subjects receiving rescue medication at Weeks 24 and 36 | 24, 36 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea Bucheon St. Mary's Hospital, Gyeonggi-do, South Korea